CLINICAL TRIAL: NCT00447915
Title: Phase II/III Clinical Study of R484iv (Ibandronic Acid) for Primary Osteoporosis - Comparative Study With Sodium Risedronate Hydrate(RIS) With Vertebral Fracture as an Index -
Brief Title: Phase II/III Clinical Study of R484iv (Ibandronic Acid) for Primary Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JA19761
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Primary Osteoporosis
MeSH Terms: interventions — Ibandronic Acid; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: ibandronic acid 0.5mg; Drug: RIS placebo; Dietary Supplement: Calcium and Vitamine D3
- 2 (Experimental)
  Interventions: Drug: RIS placebo; Drug: 1.0mg ibandronic acid; Dietary Supplement: Calcium and Vitamine D3
- 3 (Active Comparator)
  Interventions: Drug: ibandronic acid placebo; Drug: 2.5mg RIS; Dietary Supplement: Calcium and Vitamine D3

INTERVENTIONS:
Drug: ibandronic acid 0.5mg — 0.5mg(i.v.)/month for 35 months
  Arms: 1
Drug: RIS placebo — 0 mg(p.o.)/day for 36 months
  Arms: 1; 2
Drug: 1.0mg ibandronic acid — 1.0mg(i.v.)/month for 35 months
  Arms: 2
Drug: ibandronic acid placebo — 0mg(i.v.)/month for 35 months
  Arms: 3
Drug: 2.5mg RIS — 2.5 mg(p.o.)/day for 36 months
  Arms: 3
Dietary Supplement: Calcium and Vitamine D3 — Calcium 305 mg and Vitamine D3 200IU(p.o.)/day for 36 months

SUMMARY:
To evaluate the efficacy and safety of R484iv by intravenous intermittent administration to patients with primary osteoporosis in comparison with sodium risedronate hydrate (RIS) by oral administration every day. To evaluate also the dose response of R484iv.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fragile bone fracture
* Patients in whom either of study site analysis value of bone density of lumbar spine, proximal part of femur or neck of femur is less than 80% of young adult mean (YAM).
* Patients with 1 - 5 bone fractures in 4th thoracic spine (Th4) - 4th lumbar spine (L4)
* Ambulatory

Exclusion Criteria:

* Patients with disease lowering bone volume secondarily (secondary osteoporosis)
* Patients receiving at least one time of of oral bisphosphonate preparations within 6 months before the start of administration of the study drug
* Patient with disorder delaying the passage of food through esophagus

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1265 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of vertebral fracture | 36 months

SECONDARY OUTCOMES:
Change of bone density of lumbar spine and proximal part of femur from baseline | 36 months
Change of bone absorption marker from baseline | 36 months
Change of bone formation marker from baseline | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Toshitaka Nakamura, Study Chair — University of Occupational and Environment Health
Locations (4):
- Japan (4):
  - Chubu/Kansai region, Chubu/Kansai
  - Chugoku/Kyusyu region, Chugoku/Kyusyu
  - Hokkaido/Tohoku region, Hokkaido/Tohoku
  - Kanto/Koshinetsu region, Kanto/Koshinetsu